CLINICAL TRIAL: NCT01401894
Title: Pilot Study to Investigate Advanced Cancer Patient's Perspective of Their Prognosis, Goals of Treatment, and Quality of Communication With Their Oncologists
Brief Title: Perception Prognosis, Goals of Treatment, and Communication
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Director MGH BMT Survivorship Program, Massachusetts General Hospital
Other Study IDs: 10-219
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Gastric Cancer; Esophageal Cancer; Pancreatic Cancer; Liver Cancer; Biliary Cancer
Keywords: advanced cancer
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research study is to assess what the participant understands about their illness, prognosis, the goals of the cancer treatment and their communication with their oncology providers. This study will help us to figure out how the investigators can improve how other patients understand their illness and goals of treatment and help us improve communication with their doctors. This research is being done because there is not a lot of information on how much patients understand about their illness and prognosis.

DETAILED DESCRIPTION:
* Participants will be asked to answer a few basic questions regarding race, ethnicity, religion, relationship status, education, income, and living situation.
* They will then be asked to complete a questionnaire which contains questions about their mood, spirituality, quality of life and their understanding of their treatment and prognosis and their communication with their oncologist. They will complete these questionnaires in the clinic or infusion room on one of their regularly scheduled visit.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed new diagnosis of advanced gastric, esophageal, pancreatic, and hepatobiliary cancer, not being treated with curative intent.
* Planning to receive chemotherapy at Massachusetts General Hospital
* Ability to read and respond to questions in English.

Exclusion Criteria:

* Prior chemotherapy for current stage of disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a recent diagnosis of advanced gastric, esophageal, pancreatic and hepatobiliary cancer, not being treated with curative intent and receiving their cancer care at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-10; Primary Completion 2012-10 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Completion of surveys | 1 year

SECONDARY OUTCOMES:
Patients perceptions of prognosis, goals of care, and communication with providers | 1 year
Quality of end of life care | 1 year
Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States